CLINICAL TRIAL: NCT06397118
Title: Prevention of Malnutrition in Children With Sickle Cell Disease Living in Northern Nigeria
Brief Title: Prevention of Malnutrition in Children With Sickle Cell Disease
Acronym: PMC-SCD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Aminu Kano Teaching Hospital (Other); Murtala Muhammed Specialist Hospital (Other)
Responsible Party: Principal Investigator, Lauren Klein, Instructor of Pediatric Gastroenterology, Hepatology, and Nutrition, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 240090
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease; Malnutrition
Keywords: Malnutrition; Malnourishment; Undernutrition; Nutritional Deficiency; Sickle Cell Disease; Nigeria; Primary Prevention; Vitamin A; Infant and Young Child Feeding
MeSH Terms: conditions — Anemia, Sickle Cell; Malnutrition | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly allocated to intervention or control groups in a 1:1 ratio via a permuted block allocation scheme stratified by sex.
Who Masked: Outcomes Assessor
Masking Description: A trained anthropometrist will be masked to the study allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care plus Maternal Nutrition Education (Experimental): Mothers whose infants are assigned to this group will be provided individually by a community health worker during weeks 0, 8, and 16. In addition to receiving nutrition counseling, maternal nutrition education will emphasize utilizing locally available foods to enhance the nutritional well-being of young children and families, all while respecting local cultural and religious customs. To reinforce these educational messages, visual aids will be incorporated. The following educational messages will be addressed:
  1. appropriate feeding frequency
  2. dietary diversity using local foods
  3. Complementary food preparation
  4. adequate portions
  5. individualized, tailored economic education regarding the cost of purchasing foods that can fill nutrient gaps (self-efficacy)
  Interventions: Behavioral: Maternal Nutrition Education; Behavioral: Standard Care
- Standard Care Only (Active Comparator): Mothers whose infants are assigned to the control group will receive standard nutrition education from the provider at the SCD clinic during weeks 0, 8, and 16.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Maternal Nutrition Education — Community Health Worker delivered Maternal Nutrition Education
  Arms: Standard Care plus Maternal Nutrition Education
Behavioral: Standard Care — Standard care in the sickle cell disease (SCD) clinic

SUMMARY:
The investigators are studying how to prevent malnutrition in children with sickle cell disease (SCD) in northern Nigeria. Community health workers will teach mothers about nutritious local foods that might help children grow better than the usual advice from doctors. The investigators will enroll 148 children with SCD aged 6 to 18 months old. The investigators will determine if their weight and diet improve and check for low vitamin A levels. This information will help us find better ways to improve growth for children with SCD.

DETAILED DESCRIPTION:
Despite efforts to improve nutrition, 45% of under-5 mortality is at least partially attributable to malnutrition. Children with SCD have high nutrient demands and energy expenditures with a risk of impaired growth. The investigators will test the hypothesis that maternal nutrition education on locally available nutrient-dense foods will lead to improved childhood growth compared to standard pediatrician-delivered nutrition counseling. The research will involve a randomized controlled trial with 148 children aged 6 to 18 months with SCD, assessing changes in weight-for-age z-scores and dietary adequacy, as well as determining the prevalence of vitamin A deficiency. These preliminary findings will inform evidence-based interventions for the primary prevention of malnutrition (underweight and vitamin A deficiency) in children with SCD.

ELIGIBILITY:
Inclusion Criteria:

* laboratory confirmed SCD (HbSS, HbSβ0 thalassemia, or HbSC)
* aged 6 to 18 months.

Exclusion Criteria:

* severe acute malnutrition (weight-for-length z-score <-3 or mid-upper arm circumference <11.5 cm)
* diagnosis of HIV or other chronic illnesses

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in weight for the for-age z score. | 24 weeks
  Mean change in weight-for-age z score in the randomly allocated groups, standard care versus the novel maternal intervention. This is a continuous outcome where a higher z-score indicates a positive outcome.

SECONDARY OUTCOMES:
Percentage of children receiving the minimum dietary adequacy | 24 weeks
  percentage of young children with a World Health Organization-defined minimum acceptable diet based on dietary diversity and feeding frequency
Prevalence of vitamin A deficiency | 24 weeks
  Continuous unadjusted and inflammation-adjusted retinol levels and the corresponding prevalence of vitamin A deficiency

OTHER OUTCOMES:
Change in weight-for-length z-score | 24 weeks
  Mean change in weight-for-length z-score in the randomly allocated groups, standard care versus the novel maternal intervention. This is a continuous outcome where a higher z-score indicates a positive outcome.
Change in length-for-age z-score | 24 weeks
  Mean change in length-for-age z-score in the randomly allocated groups, standard care versus the novel maternal intervention. This is a continuous outcome where a higher z-score indicates a positive outcome.
Change in mid-upper arm circumference measurement | 24 weeks
  Mean change in mid-upper arm circumference measurement in the randomly allocated groups, standard care versus the novel maternal intervention. This is a continuous outcome where a mid-upper arm circumference indicates a positive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren J Klein, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wastnedge E, Waters D, Patel S, Morrison K, Goh MY, Adeloye D, Rudan I. The global burden of sickle cell disease in children under five years of age: a systematic review and meta-analysis. J Glob Health. 2018 Dec;8(2):021103. doi: 10.7189/jogh.08.021103. PMID 30574296
- [Background] GBD 2021 Sickle Cell Disease Collaborators. Global, regional, and national prevalence and mortality burden of sickle cell disease, 2000-2021: a systematic analysis from the Global Burden of Disease Study 2021. Lancet Haematol. 2023 Aug;10(8):e585-e599. doi: 10.1016/S2352-3026(23)00118-7. Epub 2023 Jun 15. PMID 37331373
- [Background] World Health Organization (WHO). Malnutrition Fact Sheets. Published 2021. Accessed June 4, 2022. https://www.who.int/news-room/fact-sheets/detail/malnutrition
- [Background] National Population Commission (NPC) [Nigeria], ICF. Nigeria Demographic and Health Survey 2018.; 2019. Accessed June 26, 2021. www.DHSprogram.com.
- [Background] Park H, Schall J, Zemel B, et al. Parameters of vitamin A (VA) status in children with sickle cell disease (SCD). The FASEB Journal. 2009;23(S1):730.5-730.5. doi:10.1096/fasebj.23.1 supplement.730.5
- [Background] Stevens GA, Bennett JE, Hennocq Q, Lu Y, De-Regil LM, Rogers L, Danaei G, Li G, White RA, Flaxman SR, Oehrle SP, Finucane MM, Guerrero R, Bhutta ZA, Then-Paulino A, Fawzi W, Black RE, Ezzati M. Trends and mortality effects of vitamin A deficiency in children in 138 low-income and middle-income countries between 1991 and 2013: a pooled analysis of population-based surveys. Lancet Glob Health. 2015 Sep;3(9):e528-36. doi: 10.1016/S2214-109X(15)00039-X. PMID 26275329
- [Background] Imdad A, Mayo-Wilson E, Herzer K, Bhutta ZA. Vitamin A supplementation for preventing morbidity and mortality in children from six months to five years of age. Cochrane Database Syst Rev. 2017 Mar 11;3(3):CD008524. doi: 10.1002/14651858.CD008524.pub3. PMID 28282701
- [Background] Thurstans S, Sessions N, Dolan C, Sadler K, Cichon B, Isanaka S, Roberfroid D, Stobaugh H, Webb P, Khara T. The relationship between wasting and stunting in young children: A systematic review. Matern Child Nutr. 2022 Jan;18(1):e13246. doi: 10.1111/mcn.13246. Epub 2021 Sep 5. PMID 34486229
- [Background] Black RE, Allen LH, Bhutta ZA, Caulfield LE, de Onis M, Ezzati M, Mathers C, Rivera J; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: global and regional exposures and health consequences. Lancet. 2008 Jan 19;371(9608):243-60. doi: 10.1016/S0140-6736(07)61690-0. No abstract available. PMID 18207566
- [Background] Klein LJ, Abdullahi SU, Gambo S, Stallings VA, Acra S, Rodeghier M, DeBaun MR. Underweight children older than 5 years with sickle cell anemia are at risk for early mortality in a low-resource setting. Blood Adv. 2023 Jun 13;7(11):2339-2346. doi: 10.1182/bloodadvances.2022008623. PMID 36383708
- [Background] Bailey J, Lelijveld N, Khara T, Dolan C, Stobaugh H, Sadler K, Lino Lako R, Briend A, Opondo C, Kerac M, Myatt M. Response to Malnutrition Treatment in Low Weight-for-Age Children: Secondary Analyses of Children 6-59 Months in the ComPAS Cluster Randomized Controlled Trial. Nutrients. 2021 Mar 24;13(4):1054. doi: 10.3390/nu13041054. PMID 33805040